CLINICAL TRIAL: NCT03062085
Title: Visual Outcome Evaluation and Genetic Analysis: Shanghai High Myopia Study
Brief Title: Shanghai High Myopia Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai High Myopia Study Group (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC-81670835
Record Dates: First submitted 2017-01-23; First posted 2017-02-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: High Myopia; Cataract; Visual Outcome; Genetic Anticipation
MeSH Terms: conditions — Cataract; Anticipation, Genetic | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples from HMC, ARC and anisometropia patients collected before the cataract surgery. Aqueous humor and capsular membranes samples from HMC, ARC and ametropic cataract patients collected during the cataract surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High myopic cataract group: Cataract patients with high myopia.
  Interventions: Other: Cataract
- Age-related cataract group: Age-related cataract patients.
  Interventions: Other: Cataract
- Ametropic cataract group: Cataract patients with ametropia.
  Interventions: Other: Cataract

INTERVENTIONS:
Other: Cataract — The genetic and environmental factors concerning to the pathogenesis of cataract in the three groups.

SUMMARY:
The purpose of this study is to evaluate the long-term visual outcome of the cataract surgery using a large-scale and comprehensive database of high myopic cataract and age-related cataract patients. The investigators will further investigate into the various genetic and environmental factors that may contribute to the pathogenesis of high myopic cataract.

DETAILED DESCRIPTION:
High myopic cataract (HMC) has become a major high-risky type of cataract in China, which accounts for nearly 30% of cataract in recent years. Compared to age-related cataract, HMC is characterized with earlier onset, severer lens opacities, higher incidence of vitreoretinopathy and postoperative complications compared to age-related cataract(ARC).

The main purpose of this study is to evaluate the long-term visual outcome of the cataract surgery using a large-scale and comprehensive database of high myopic cataract, when compared to those age-matched ARC patients.

On the other hand, due to the lack of research in the pathogenesis of HMC, it is difficult for the investigators to precisely evaluate its risk and prognosis, and to improve its prevention and treatment. The previous study of investigators majored in a large-sample analysis on the clinical features and related genes of HMC. After preliminary screening, eight genes were selected for further investigation: 1) genes related to pathogenesis of HMC: CRYAA/ GSTP1/ TXNRD2;2) genes related to vitreoretinopathy: MCP1/ VEGFA/ CFH; 3) genes related to postoperative complications: TGFB2/ CERS2. In the present study, in order to establish a risk model of HMC from the aspect of precision medicine, the investigators are preparing to set up a comprehensive clinical database for further sequencing of selected genes (including exons, promoters, 5' UTR and 3' UTR sequences) on a large scale, to intensively investigate into the sites and functions of single nucleotide polymorphism (SNP) correlated with clinical features of HMC.

The research aim to evaluate the long-term visual outcome of the cataract surgery using a large-scale and comprehensive database of high myopic cataract, to thoroughly illustrate the influence of HMC-related genes to its prognosis and to elucidate the pathogenesis of HMC, for further promotion in the disease prevention and prognosis as well.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cataract
* Must be able to cooperate with the ophthalmic examination

Exclusion Criteria:

* Clinical diagnosis of mental illness
* Mentally disabled

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract patients who will undergo cataract surgery in Eye and ENT Hospital of Fudan University.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the clinical phenotypes and visual outcomes of high myopic cataract patients | Follow-up until five years after surgery
  Cataract type and severity of high myopic cataract patients are evaluated using LOCSIII grading system. Visual outcomes are also evaluated including visual acuity with or without correction, intraocular pressure, fundus function, contrast sensitivity and other visual outcome measurements.
Differences in the clinical phenotypes and visual outcomes of age-related cataract patients | Follow-up until five years after surgery
  Cataract type and severity of age-related cataract patients are evaluated using LOCSIII grading system. Visual outcomes are also evaluated including visual acuity with or without correction, intraocular pressure, fundus function, contrast sensitivity and other visual outcome measurements.
Differences in the clinical phenotypes and visual outcomes of ametropic cataract patients | Follow-up until five years after surgery
  Cataract type and severity of ametropic cataract patients are evaluated using LOCSIII grading system. Visual outcomes are also evaluated including visual acuity with or without correction, intraocular pressure, fundus function, contrast sensitivity and other visual outcome measurements.

SECONDARY OUTCOMES:
Genetic diversity based on biological specimen samples of three groups | Analyzed within six months after surgery
  Sequencing of selected genes (including exons, promoters, 5' UTR and 3' UTR sequences) on a large scale to intensively investigate into the sites and functions of single nucleotide polymorphism (SNP) correlated with clinical features of HMC, compared to age-related cataract and ametropic cataract patients.

OTHER OUTCOMES:
Difference in the surgical procedure of three groups | Recorded on the surgery day for further analysis
  To compare the difference in the surgical procedure of three groups.
Difference in the Diagnostic test of three groups | Recorded before the surgery day for further analysis
  To compare the difference in the diagnostic test of three groups.
Difference in the complications of the cataract surgery of three groups | Follow-up until five years after surgery
  To compare the prevalence of complications of the cataract surgery in HMC,ARC and ametropic cataract patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, M.D., Study Chair — Eye and ENT Hospital of Fudan University; Xiangjia Zhu, M.D., Study Director — Eye and ENT Hospital of Fudan University; Keke Zhang, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Wenwen He, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Yu Du, B.S., Principal Investigator — Eye and ENT Hospital of Fudan University; Yinglei Zhang, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Zhennan Zhao, Ph.D., Principal Investigator — Eye and ENT Hospital of Fudan University; Ruiqi Chang, B.S., Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Derived] Zhang Y, Zhang S, Zhang K, Lu Y, Zhu X. Characteristics of the Corneal Endothelium in Elderly Adults with High Myopia. Phenomics. 2025 Jan 27;4(6):562-569. doi: 10.1007/s43657-024-00186-6. eCollection 2024 Dec. PMID 40061825
- [Derived] Hu X, Qi J, Cheng K, He W, Zhang K, Zhao C, Lu Y, Zhu X. Effectiveness of prophylactic capsular tension ring implantation during cataract surgery in highly myopic eyes. J Cataract Refract Surg. 2024 Oct 1;50(10):1030-1036. doi: 10.1097/j.jcrs.0000000000001495. PMID 39313860
- [Derived] He W, Wei L, Liu S, Huang Z, Qi J, Zhang K, Meng J, Du Y, Lu Y, Zhu X. Role of Optic Nerve Head Characteristics in Predicting Intraocular Pressure Spikes after Cataract Surgery in Highly Myopic Eyes. Ophthalmol Ther. 2023 Aug;12(4):2023-2033. doi: 10.1007/s40123-023-00714-z. Epub 2023 May 13. PMID 37178442
- [Derived] He W, Cheng K, Zhao L, Liu S, Huang Z, Zhang K, Du Y, Zhou X, Lu Y, Zhu X. Long-Term Outcomes of Posterior Capsular Opacification in Highly Myopic Eyes and Its Influencing Factors. Ophthalmol Ther. 2023 Aug;12(4):1881-1891. doi: 10.1007/s40123-023-00711-2. Epub 2023 May 3. PMID 37138195
- [Derived] Meng J, Chen Y, Cheng K, Qi J, Du Y, Yao Y, He W, Zhang K, Lu Y, Zhu X. LONG-TERM PROGRESSION PATTERN OF MYOPIC TRACTIONAL MACULOPATHY: Outcomes and Risk Factors. Retina. 2023 Jul 1;43(7):1189-1197. doi: 10.1097/IAE.0000000000003791. PMID 36977327
- [Derived] Lu Q, He W, Qian D, Lu Y, Zhu X. Measurement of crystalline lens tilt in high myopic eyes before cataract surgery using swept-source optical coherence tomography. Eye Vis (Lond). 2020 Mar 6;7:14. doi: 10.1186/s40662-020-00176-5. eCollection 2020. PMID 32161773